CLINICAL TRIAL: NCT00578344
Title: Allogeneic Bone Marrow Transplantation From HLA Identical Related Donors for Patients With Hemoglobinopathies: Hemoglobin SS, Hemoglobin SC, or Hemoglobin SB0/+ Thalassemia
Brief Title: Bone Marrow Transplantation, Hemoglobinopathies, SCALLOP
Acronym: SCALLOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to no new subject enrollment during the last 3 year period.
Sponsor: Tami D. John (Other)
Collaborators: Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Tami D. John, Assistant Professor, Pediatrics-Hema & Oncology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16447-SCALLOP; SCALLOP (Other: Baylor College of Medicine)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Sickle Cell Disease; Hemoglobin SC
Keywords: Sickle Cell Disease; SCD; Hemoglobin SS; Hemoglobin SC; Hemoglobin Sb0/+; HLA genotype; Severe anemia; Transfusion therapy
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease; Anemia | interventions — Busulfan; Alemtuzumab; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic BMT/SCT Transplant (Experimental): Busulfan, Campath 1H, Cyclophosphamide and MESNA:
  Bone marrow infusion with pre-meds as per SOPs to take place on Day 0.
  Bone marrow dose: To ensure the probability for bone marrow engraftment, 4 x 10^8 nucleated cells/kg patient weight will be the target at donor bone marrow harvest.
  Interventions: Drug: Busulfan; Biological: Campath 1H; Drug: Cyclophosphamide and MESNA

INTERVENTIONS:
Drug: Busulfan — Starting Day -9 / Busulfan 4.0 mg/kg/day IV divided into four doses daily for four days; total dose = 16 mg/kg.
  Other Names: Myleran
Biological: Campath 1H — Day -5 through Day -2; Campath-1H dosed as per institutional guidelines.
Drug: Cyclophosphamide and MESNA — Day -5 through Day -2; Cyclophosphamide 50 mg/kg + MESNA.
  Other Names: CTX

SUMMARY:
Patients are being asked to participate in this study because they have severe sickle cell anemia (SCD) with or without the beta thalassemia trait. Sickle cell anemia is an illness where the red blood cells change shape and can clog up blood vessels. This keeps the body from getting the oxygen it needs. Thalassemia is when the body does not make enough hemoglobin, something that helps the oxygen get to the places it needs to go in the body. The patient may or may not need to get regular blood transfusions (getting more blood) to improve their quality of life (feel better) and prevent organ damage (problems with the brain, heart, lung, kidney, and gonad, for example.). The transfusions can also cause problems, including iron overload (too much iron in the blood), which can be fatal (patients can die) without regular deferoxamine shots. Even with the best usual treatments, people with thalassemia or SCD die sooner. There is no proven cure.

We would like to treat patients using bone marrow transplantation, a treatment that has been used for people with SCD. The transplant uses healthy "matched" bone marrow. This comes from a brother or sister who does not have sickle cell disease or severe thalassemia. If the treatment works, the sickle cell disease or thalassemia may be cured. This treatment has been used to treat patients with sickle cell disease or thalassemia. It has worked in most cases. We hope, but cannot promise, that the transplanted marrow will make healthy cells, and patients will not have sickle cell disease or severe thalassemia anymore.

We do not know what effect this treatment will have on the damage that has already been done by the disease. Finding that out is the main reason for this study. Currently, very little has been reported about organ function after bone marrow transplants in patients with sickle cell anemia.

DETAILED DESCRIPTION:
Prior to any bone marrow transplant, we will need patients to:

* Answer questions about their medical history;
* Undergo a physical examination;
* Have tests done to see how well the lungs are working;
* Have a chest x-ray;
* Have an EKG to look at the heart;
* Have an MRI & MRA (Magnetic Resonance Angiography, which looks at the blood vessels and the blood flowing through them). These 2 tests will look to see if the patient has had any strokes;
* Have a PET scan to look at the head and body;
* Have a liver biopsy to determine if the liver has been damaged (which can happen from iron overload that happens after many transfusions). Too much liver damage would mean a transplant cannot be done.

For the liver biopsy, the skin is numbed with medicine, and a special needle goes into the liver. The needle removes a very small piece of the liver (tissue). The tissue is taken and examined.

Also, about 30 cc (2 tablespoons) of blood will be drawn to test the blood for viruses, including HIV (the virus that causes AIDS). If the HIV test is positive, a transplant will not be done because it would be too dangerous for the patient.

At least 2 weeks before the bone marrow infusion, the patient will be immunized with Prevnar 7. Prevnar 7 is a vaccine that is used in children to protect against some types of bacteria called Streptococcus pneumoniae, which can cause the lung infection called pneumonia. People with Sickle Cell anemia are at a higher risk of dying from an infection from this type of bacteria. Although children are regularly given the Prevnar 7 vaccine, it is not common to test a child's immune response to the vaccine. In this study, we will check the immune system's response to the vaccine by drawing an extra 3 mL (less than 1 teaspoon) of blood 3 weeks after the patient gets the Prevnar 7 vaccine.

Just before the bone marrow transplant, we must kill the cells in the bone marrow that make the abnormal red blood cells found in patients with severe thalassemia or sickle cell disease. We will do this by using 3 drugs: busulfan, cyclophosphamide, and campath-1H. Campath-1H is used to prevent the body from rejecting or refusing to let the donor blood cells grow in the body. MESNA is given with the cyclophosphamide to prevent kidney damage. Methotrexate and cyclosporin are also given to prevent graft-versus-host disease (GVHD); methylprednisolone will be given after the bone marrow infusion if the patient develops GVHD. A drug will also be given to prevent seizures (either dilantin or lorazepam).

Graft-versus-host disease (GVHD) is a possible side-effect of the transplant. In GVHD, some cells in the donor marrow attack cells in the patient's body. This causes skin, liver, and bowel problems, and may damage other parts of the body. Often, these problems are fairly mild, but they can be severe or even cause death. Severe GVHD is likely to occur in about 10% of patients.

After the patient gets the drug treatment, they will be given bone marrow from a brother or sister who has healthy bone marrow that matches the patients. The healthy bone marrow will be put into a vein (given IV) in the same way that blood transfusions are given. The marrow cells then travel to the right places in the body, where they should grow and make new normal blood cells.

This is the treatment schedule:

Protocol Day & Treatment:

14 or more days before the bone marrow infusion -- Prevnar 7 vaccine

10 days before the bone marrow infusion -- Begin Dilantin or Lorazepam (to prevent seizures)

9 days before the bone marrow infusion -- Busulfan

8 days before the bone marrow infusion -- Busulfan

7 days before the bone marrow infusion -- Busulfan

6 days before the bone marrow infusion -- Busulfan

5 days before the bone marrow infusion -- Campath 1H, Cyclophosphamide, and MESNA

4 days before the bone marrow infusion -- Campath 1H, Cyclophosphamide, and MESNA

3 days before the bone marrow infusion -- Campath 1H, Cyclophosphamide, and MESNA

2 days before the bone marrow infusion -- Campath 1H, Cyclophosphamide, MESNA, and cyclosporin

1 day before the bone marrow infusion -- DAY OF REST

Day "0" -- bone marrow infusion given

1 day after the bone marrow infusion -- Methotrexate

3 days after the bone marrow infusion -- Methotrexate

6 days after the bone marrow infusion -- Methotrexate

11 days after the bone marrow infusion -- Methotrexate

After transplant, Filgrastrim, a growth hormone for the bone marrow, may be given intravenously (through a vein), if medically necessary.

Sometimes, the donor's bone marrow does not grow. Then, the patient would be without working bone marrow cells. So that we will be ready to treat this problem if it happens, we will take bone marrow from the hip bone before the patient gets the drug treatment. The patient will be asleep (sedated) when the marrow is taken, and they will be given medicine for any pain they have afterwards. This bone marrow will be frozen and stored or preserved. If the donor bone marrow does not grow, we will thaw the stored marrow and put it back into the body. This stored bone marrow should grow and produce working blood cells. If the stored bone marrow must be given back, the disease will not be cured.

To tell whether the transplant has worked or "engrafted", we will take samples of bone marrow (bone marrow aspirate). We will do this 3 weeks after the transplant to make sure the new cells are beginning to grow. We will take another marrow sample at 3 months after the transplant. We want to make sure the new cells are still growing. This test will take about 30 to 45 minutes. Because this test is painful, the patient will be given pain medicine before, during, and after the test.

The patient will need to be in the hospital for at least 3 weeks after the transplant to make sure the transplant has engrafted. We will do several tests (of the lung, kidney, and liver) before and after the bone marrow transplant. We want to find out how much the treatment has helped the patient and how much it might help other patients. Most tests will be done every week for 4 months and at each visit to the hospital. Also, we will be looking at the immune function. To do this, we will take about 8 ml (less than 2 teaspoonful) at 6 months, 1 year, and 2 years after the transplant. When possible, we will take the blood from an IV line that the patient already has. However, at times we will have to draw the blood with another needle stick. A total amount of 200 mL (about 13 tablespoons) of blood will be collected from the patient during the entire study.

After 4 months, if the patient's health is good, they will not need to come to the hospital so often. The visits to the doctor should be more like they were before the bone marrow transplant. Since problems may happen months after the transplant and this is a new way to treat sickle cell disease and thalassemia the patient will need to have exams and blood tests done every few months during the first and second years after their transplant. After that, if all is well, the patient will need to be examined and have blood tests 4 times a year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a related HLA genotype identical donor and hemoglobin SS, hemoglobin SC, or hemoglobin Sb0/+ and at least one of the following conditions:

   1. Previous central nervous system vaso-occlusive episode with or without residual neurologic findings, or has an abnormal transcranial doppler exam without neurologic findings, or abnormal MRI/MRA of the brain with or without neurologic findings;
   2. Frequent painful vaso-occlusive episodes which significantly interfere with normal life activities and which necessitate chronic transfusion therapy;
   3. Recurrent SCD chest syndrome events, which necessitate chronic transfusion therapy;
   4. Severe anemia which prevents acceptable quality of life and necessitates chronic transfusion therapy;
   5. Any of the above symptoms in which the patient is not undergoing chronic transfusion therapy;
   6. The patient is undergoing chronic transfusion therapy for symptoms other than those listed and which significantly interferes with normal life activities;
   7. Failed hydroxyurea therapy;
   8. Indication of pulmonary hypertension on 2 separate echocardiogram examinations;
   9. Patients who plan to return to resource poor areas/countries.
2. Between the ages of birth and 40 years.
3. Women of childbearing potential must have a negative pregnancy test.

EXCLUSION CRITERIA:

1. Patient with biopsy proven chronic active hepatitis or fibrosis with portal bridging.
2. Patient with SCD chronic lung disease > stage 3 (see Appendix 1).
3. Patient with severe renal dysfunction defined as creatinine clearance < 40 mL/min/1.73 M^2.
4. Patient with severe cardiac dysfunction defined as echocardiogram shortening fraction < 25% or NYHA class III or IV.
5. Patient with HIV infection.
6. Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplantation.
7. Patient or patient's guardian(s) unable to understand the nature and risks inherent in the BMT process.
8. Pregnant/lactating women and those unwilling to use acceptable contraception will be excluded.
9. Patient or patient's guardian who have not signed an informed consent.

NOTE: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CAGT Protocol Review Committee and the FDA reviewer.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2005-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tami John, MD, Study Director — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic BMT/SCT Transplant: Busulfan, Campath 1H, Cyclophosphamide and MESNA:
  Bone marrow infusion with pre-meds as per SOPs to take place on Day 0.
  Bone marrow dose: To ensure the probability for bone marrow engraftment, 4 x 10^8 nucleated cells/kg patient weight will be the target at donor bone marrow harvest.
  Busulfan: Starting Day -9 / Busulfan 4.0 mg/kg/day IV divided into four doses daily for four days; total dose = 16 mg/kg.
  Campath 1H: Day -5 through Day -2; Campath-1H dosed as per institutional guidelines.
  Cyclophosphamide and MESNA: Day -5 through Day -2; Cyclophosphamide 50 mg/kg + MESNA.
Period: Overall Study
Arm/Group | Allogeneic BMT/SCT Transplant
Started | 8
Completed | 6
Not Completed | 2
Not completed — Insurance problems | 1
Not completed — Graft failure | 1

BASELINE CHARACTERISTICS:
Population: All participants underwent allogeneic bone marrow transplantation from human leukocyte antigen (HLA) identical related donors with hemoglobinopathies.
Arm/Group | Allogeneic BMT/SCT Transplant
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 8.5 [4 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Evidence of Recovery of Organ Function Measured Via MRI or PET Scan.
Description: Assess Number of participants that recovered organ function diagnosed with sickle cell disease (SCD) or sickle hemoglobin variants after undergoing allogeneic SCT/BMT from HLA genotype identical donors.
Time Frame: One year
Population: Out of eight participants who underwent bone marrow transplant, six participants with positron emission tomography (PET) or magnetic resonance imaging (MRI) at the time of assessment were included in the analysis. The other two were inevaluable due to graft failure or no PET or MRI at the time of assessment. Data were collected at 1 year only.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic BMT/SCT Transplant
Number analyzed (Participants) | 6
Participants
  Stable | 4
  Progressive | 2

2. Primary Outcome: Number of Participants With Pre and Post Transplant PET Scan to Assess Organ Recovery Based on Rate of Acquisition.
Description: Number of participants that did or did not have pre- and post- PET scans.
Time Frame: One year
Population: All participants who underwent allogeneic bone marrow transplantation from human leukocyte antigen (HLA) identical related donors with hemoglobinopathies were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic BMT/SCT Transplant
Number analyzed (Participants) | 8
Participants
  No pre and post PET scan | 6
  Pre and post PET scan | 2

3. Primary Outcome: Number of Participants With Immune Response to Immunization After BMT in Participants With SCD, Hemoglobin SC, or Hemoglobin Sb0/+.
Description: Vaccine response will be measured via a humoral immunity panel evaluating streptococcus pneumonia IgG antibodies (microgram/mL). Panels are obtained pre and 1+ month post vaccination. Standard recommendations define a normal responder as having >4 fold increase in antibody level in 50-70% of the serotypes found in the vaccine.
Time Frame: up to 12 months
Population: Out of eight participants who underwent bone marrow transplant, seven participants engrafted were included in the analysis. The other participant was excluded because he/she did not engraft and received a second transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic BMT/SCT Transplant
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: Primary BMT studies have a critical toxicity period of 30 days after BMT day 0. During the critical toxicity period the most severe grade of all AE's is captured. Grade 1 and 2 AEs, hematological toxicities, and fevers are excluded. Serious Adverse Events/Unanticipated Problems are reported (excluding hematological toxicities and fevers) until 100 days after BMT day 0.
Description: All adverse events were collected using CTCAE 2.0 for the study. For reporting purpose, adverse event terms were converted using CTCAE v4.0.
Arm/Group | Allogeneic BMT/SCT Transplant
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic BMT/SCT Transplant (N=8)
Catheter-related infection (Infections and infestations) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic BMT/SCT Transplant (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (8)
Blood bilirubin increased (Investigations) | 1 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders - Other: Prolonged QTc interval (QTc > 0.48 seconds) (Cardiac disorders) | 1 (1)
Cardiac disorders - Other: Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (1)
Catheter-related infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
GGT increased (Investigations) | 1 (2)
Hallucinations (Psychiatric disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other: BK viremia (Infections and infestations) | 1 (1)
Infections and infestations - Other: Candida Albicans in tongue culture (Infections and infestations) | 1 (1)
Infections and infestations - Other: Parainfluenza 3 respiratory infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (6)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT00578344/Prot_SAP_000.pdf